CLINICAL TRIAL: NCT01689701
Title: Efficacy and Safety of Hizikia Fusiformis Extract in Subjects Showing Erosive Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PKU-EG-ECKL
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Erosive Gastritis
Keywords: Erosive Gastritis; Hizikia Fusiformis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hizikia Fusiformis extract (Experimental)
  Interventions: Dietary Supplement: Hizikia Fusiformis extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hizikia Fusiformis extract — Hizikia Fusiformis extract(1.3g/d)
  Arms: Hizikia Fusiformis extract
Dietary Supplement: Placebo — Placebo(1.3g/d)
  Arms: Placebo

SUMMARY:
The investigators performed a double-blind parallel study in a group of Subjects Showing Erosive Gastritis who were given Hizikia Fusiformis Extract over a period of 4 weeks. Endoscopic observations were performed before and 4 weeks after the treatment, and the cure and improvement rates were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-70 years old
* Subjects Showing Erosive Gastritis (endoscopy)
* Able to give informed consent

Exclusion Criteria:

* Diagnosed of gastrointestinal disease such as ulcer, cancer within 1 months
* Allergic or hypersensitive to any of the ingredients in the test products
* History of disease that could interfere with the test products or impede their absorption, such as gastrointestinal disease or gastrointestinal surgery
* Taken antibiotics and stomach medicines such as steroid, bismuth compound and proton pump inhibitor within 1 months
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Wook Kim, MD, Principal Investigator — Chonbuk National University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study subjects were recruited from Clinical Trial Center for Functional Food in Chonbuk National University Hospital during the 2011. Only those subjects who were Subjects Showing Erosive Gastritis and were not diagnosed with any disease were included in this study.
Pre-assignment Details: Among the 79 subjets screened, 25 subjects had endoscopy and/or laboratory tests results that were in the exclusion criteria category, hence they were excluded from the study.
Groups:
- Hizikia Fusiformis Extract: Hizikia Fusiformis extract(1.3g/d) for 12weeks
  Hizikia Fusiformis extract: Hizikia Fusiformis by Ethanol and extracted with concentrated
- Placebo: Placebo(1.3g/day) for 4weeks
  Placebo : Amount and calorie of placebo are same with Hizikia Fusiformis extract.
Period: Overall Study
Arm/Group | Hizikia Fusiformis Extract | Placebo
Started | 27 | 27
Completed | 22 | 21
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hizikia Fusiformis Extract | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.9) | 38.7 (10.0) | 38.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Changes in Erosions
Description: Erosions was measured in study visit 1(0 week) and visit 3(4 week). Gastric erosion occurs when the mucous membrane lining the stomach becomes inflamed.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: erosions
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
erosions
  Pre | 4.36 (2.48) | 3.38 (2.89)
  Post | 2.32 (2.10) | 2.43 (3.28)

2. Primary Outcome: Changes in Score of Erosions
Description: Score of erosions(score 1-4) was measured in study visit 1(0 week) and visit 3(4 week).
  Score of erosions is assigned a score of between 1 (Erosion = 0) to 4 (Erosion ≥ 6) and summed to form a score ranging from 1 (best) to 4 (worst).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
Scores on a scale
  Pre | 3.00 (0.76) | 2.71 (0.78)
  Post | 2.23 (0.92) | 2.05 (1.12)

3. Secondary Outcome: Changes in Subjects' Symptoms Total Score
Description: Subjects' symptoms total score(score 0-24) was measured in study visit 1(0 week) and visit 3(4 week).
  The original index consists of 8 Questions. Individual question response is assigned a score of between 0 (none) to 3 (moderate) and summed to form a score ranging from 0 (best) to 24 (worst).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
Units on a scale
  Pre | 2.77 (2.56) | 3.90 (4.15)
  Post | 2.77 (3.18) | 2.57 (3.37)

4. Secondary Outcome: Changes in Gastrin
Description: Gastrin was measured in study visit 1(0 week) and visit 3(4 week).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
pg/ml
  Pre | 37.36 (16.43) | 36.44 (16.88)
  Post | 32.05 (15.27) | 27.61 (10.86)

5. Secondary Outcome: Changes in PepsinogenⅠ
Description: PepsinogenⅠ was measured in study visit 1(0 week) and visit 3(4 week).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
ng/mL
  Pre | 50.15 (14.78) | 54.72 (16.24)
  Post | 55.28 (19.08) | 57.96 (19.42)

6. Secondary Outcome: Changes in PepsinogenⅡ
Description: PepsinogenⅡ was measured in study visit 1(0 week) and visit 3(4 week).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
ng/ml
  Pre | 13.40 (8.38) | 12.65 (7.46)
  Post | 15.39 (10.16) | 13.66 (8.09)

7. Secondary Outcome: Changes in Pepsinogen Ⅰ/Ⅱ Ratio
Description: Pepsinogen Ⅰ/Ⅱ ratio was measured in study visit 1(0 week) and visit 3(4 week).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Pre | 4.66 (1.86) | 5.17 (1.83)
  Post | 4.56 (1.84) | 5.07 (1.73)

8. Secondary Outcome: Changes in Hs-CRP(High Sensitivity C-reactive Protein)
Description: Hs-CRP(High Sensitivity C-reactive Protein) was measured in study visit 1(0 week) and visit 3(4 week).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Hizikia Fusiformis Extract | Placebo
Number analyzed (Participants) | 22 | 21
mg/L
  Pre | 0.63 (1.24) | 0.16 (0.19)
  Post | 0.23 (0.4) | 0.75 (2.01)

ADVERSE EVENTS:
Arm/Group | Hizikia Fusiformis Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No